CLINICAL TRIAL: NCT01047930
Title: The Effect of Exercise on Acute Nicotine Withdrawal: Human Study
Brief Title: The Effect of Exercise on Acute Nicotine Withdrawal
Acronym: NicEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Isabella Soreca, Assistant Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO09060305; 1R01DA027508-01 (NIH)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Nicotine Dependence; Smoking; Sleep Disorders, Intrinsic
Keywords: Insomnia; Smoking; Cue reactivity; Exercise timing; Acute nicotine withdrawal; Mood disturbances; Smoking abstinence; Exercise intensity; Altered sleep; Exercise duration; Nonpharmacologic behavioral treatment; Smoking cessation; Exercise Test; Polysomnography
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Sleep Disorders, Intrinsic; Sleep Initiation and Maintenance Disorders; Smoking Cessation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AM-Ex; PM-Ex; C (Other): within subject design, with each participant receiving all three conditions
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Each 3-day experimental period will include one of the following conditions:
  1. Morning exercise - subject will exercise on each of the three mornings in the sleep laboratory, starting 30 minutes after their habitual rise-time;
  2. Evening exercise - subject will start exercise 4 hours before their habitual bedtime on each of the three evenings;
  3. No exercise - subject will watch television or read and they will be required to remain sedentary.

SUMMARY:
The primary aim of this project is to test the effect of exercise on acute nicotine withdrawal. Acute nicotine withdrawal is characterized by a complex array of symptoms associated with increased risk of relapse among individuals attempting smoking cessation. The available remedies do not target all aspects of withdrawal. For example, pharmacologic treatments reduce withdrawal-based craving, but have no effect on cue-related craving, altered sleep, and mood disturbances during withdrawal. Therefore, non-pharmacologic behavioral techniques with the potential to attenuate persistent withdrawal symptoms are needed. We hypothesized that exercise can be a valid non-pharmacologic strategy to improve these domains.

DETAILED DESCRIPTION:
The goal of the proposed work is to test: 1) the effects of exercise on mood, objective measures of sleep, and cue reactivity; 2) the effects of exercise at a given intensity and duration, after a short (few hours) and more prolonged (24 to 72 hours) abstinence from smoking; and 3) the effects of exercising in the morning versus exercising in the evening on the proposed outcome domains. We plan to implement a within-subject design that will allow us to collect measures for each subject aged 18 to 45 in four different conditions: 1) ad libitum smoking; 2) evening exercise after 2 to 72 hours of abstinence; 3) morning exercise after 2 to 72 hours of abstinence; and 4) no exercise after 2 to 72 hours of abstinence. Exercise will be conducted at a fixed and monitored dose and duration. By collecting morning and evening measures of withdrawal symptoms and cue reactivity, we will also test whether the effects of exercise in reducing withdrawal symptoms and cue reactivity will show a prolonged effect beyond the minutes/hours immediately after the exercise bout. We also hypothesize that the timing of exercise may have differential effects on different aspect of withdrawal. The proposed work will allow us to examine the extent to which exercise, a promising nonpharmacologic behavioral treatment method, can attenuate key symptoms of withdrawal recognized to impede abstinence efforts. A better understanding of these effects will allow us to implement exercise at the time of day that may be more troublesome for the individual attempting to quit. The development of new behavioral methods for attenuating withdrawal symptoms will be directly transferable to smoking cessation treatments aimed at reducing withdrawal symptoms and aiding efforts to avoid relapse after quitting smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Not regularly exercising, defined as exercising fewer than three times per week and for no more than 20 minutes each time
* Free of medical illnesses (need to be cleared by a physician as able to exercise at 60% maximum heart rate (MHR))
* Currently meeting DSM-IV criteria for nicotine dependence (No Current or Past history of any other psychiatric disorder)
* Regularly smoking at least 08 cigarettes per day for at least 12 consecutive months, not attempted to quit smoking in the previous month, and not currently taking medication for smoking cessation
* Currently displaying carbon monoxide breath readings >10 and urine cotinine levels >3
* Habitual bedtime between 9:30 p.m. and 1:30 a.m.
* Body Mass Index (BMI) less than 40.

Exclusion Criteria:

* Unable to exercise
* Currently diagnosed or treated for any psychiatric disorder; treatment with psychotropic medication will be considered on a case by case basis
* History or active treatment or any treatment in past year for any mood or psychotic disorder
* Current or past diagnosis of a sleep disorder
* Currently taking sleep medications or other medications known to alter sleep architecture
* Currently doing shift work or working at night
* History of travel across time zones in the past month
* For women of child bearing potential: pregnant or actively trying to become pregnant
* Parent of a child under two years of age
* Diagnosis of Sleep Apnea

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Primary variables of interest are self-rating score of mood, objective measures of sleep latency and WASO, subjective ratings of craving, and cardiovascular reactivity including blood pressure and heart rate reactivity during cue reactivity. | 7/2013

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Soreca, M.D., Principal Investigator — University of Pittsburgh Medical Center, Western Psychiatric Institute and Clinic
Locations (1):
- University of Pittsburgh Medical Center, Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] al'Absi M, Amunrud T, Wittmers LE. Psychophysiological effects of nicotine abstinence and behavioral challenges in habitual smokers. Pharmacol Biochem Behav. 2002 Jun;72(3):707-16. doi: 10.1016/s0091-3057(02)00739-6. PMID 12175468
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, fourth edition. American Psychiatric Association, Washington, DC, 1994
- [Background] Anton MM, Cortez-Cooper MY, DeVan AE, Neidre DB, Cook JN, Tanaka H. Resistance training increases basal limb blood flow and vascular conductance in aging humans. J Appl Physiol (1985). 2006 Nov;101(5):1351-5. doi: 10.1152/japplphysiol.00497.2006. Epub 2006 Jul 13. PMID 16840576
- [Background] Audrain-McGovern J, Rodriguez D, Moss HB. Smoking progression and physical activity. Cancer Epidemiol Biomarkers Prev. 2003 Nov;12(11 Pt 1):1121-9. PMID 14652270
- [Background] Benowitz NL. Neurobiology of nicotine addiction: implications for smoking cessation treatment. Am J Med. 2008 Apr;121(4 Suppl 1):S3-10. doi: 10.1016/j.amjmed.2008.01.015. PMID 18342164
- [Background] Biddle SJH, Fox KR, Boutcher SH (Eds): Physical activity and psychological well-being. Routledge, New York, NY, 2000.
- [Background] Blakesley RE, Mazumdar S, Dew MA, Houck PR, Tang G, Reynolds CF 3rd, Butters MA. Comparisons of methods for multiple hypothesis testing in neuropsychological research. Neuropsychology. 2009 Mar;23(2):255-64. doi: 10.1037/a0012850. PMID 19254098
- [Background] Chen X, Wei L. A comparison of recent methods for the analysis of small-sample cross-over studies. Stat Med. 2003 Sep 30;22(18):2821-33. doi: 10.1002/sim.1537. PMID 12953282
- [Background] Ekkekakis P. Pleasure and displeasure from the body: Perspectives from exercise. Cogn Emot. 2003 Mar;17(2):213-239. doi: 10.1080/02699930302292. PMID 29715726
- [Background] Ekkekakis P, Hall EE, Petruzzello SJ. The relationship between exercise intensity and affective responses demystified: to crack the 40-year-old nut, replace the 40-year-old nutcracker! Ann Behav Med. 2008 Apr;35(2):136-49. doi: 10.1007/s12160-008-9025-z. Epub 2008 Mar 28. PMID 18369689
- [Background] Ekkekakis P, Hall EE, Petruzzello SJ. Variation and homogeneity in affective responses to physical activity of varying intensities: an alternative perspective on dose-response based on evolutionary considerations. J Sports Sci. 2005 May;23(5):477-500. doi: 10.1080/02640410400021492. PMID 16194996
- [Background] Fox KR. The influence of physical activity on mental well-being. Public Health Nutr. 1999 Sep;2(3A):411-8. doi: 10.1017/s1368980099000567. PMID 10610081
- [Background] Grove RJ, Wilkinson A, Dawson B, Eastwood P, Heard P: Effects of exercise on subjective aspects of sleep during tobacco withdrawal. Aust Psychol 41:69-76, 2006.
- [Background] Hughes JR. Effects of abstinence from tobacco: valid symptoms and time course. Nicotine Tob Res. 2007 Mar;9(3):315-27. doi: 10.1080/14622200701188919. PMID 17365764
- [Background] Johnson RA, Wichern DW: Applied Multivariate Statistical Analysis, 5th edition. Prentice Hall, Upper Saddle River, NJ, 2002.
- [Background] Kenny PJ, Markou A. Neurobiology of the nicotine withdrawal syndrome. Pharmacol Biochem Behav. 2001 Dec;70(4):531-49. doi: 10.1016/s0091-3057(01)00651-7. PMID 11796152
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Netz Y, Zach S, Taffe JR, Guthrie J, Dennerstein L. Habitual physical activity is a meaningful predictor of well-being in mid-life women: a longitudinal analysis. Climacteric. 2008 Aug;11(4):337-44. doi: 10.1080/13697130802239083. PMID 18645700
- [Background] Nides MA, Rakos RF, Gonzales D, Murray RP, Tashkin DP, Bjornson-Benson WM, Lindgren P, Connett JE. Predictors of initial smoking cessation and relapse through the first 2 years of the Lung Health Study. J Consult Clin Psychol. 1995 Feb;63(1):60-9. doi: 10.1037//0022-006x.63.1.60. PMID 7896992
- [Background] Ortega FB, Ruiz JR, Castillo MJ, Sjostrom M. Physical fitness in childhood and adolescence: a powerful marker of health. Int J Obes (Lond). 2008 Jan;32(1):1-11. doi: 10.1038/sj.ijo.0803774. Epub 2007 Dec 4. PMID 18043605
- [Background] Paavola M, Vartiainen E, Puska P. Smoking cessation between teenage years and adulthood. Health Educ Res. 2001 Feb;16(1):49-57. doi: 10.1093/her/16.1.49. PMID 11252283
- [Background] Piasecki TM, Fiore MC, Baker TB. Profiles in discouragement: two studies of variability in the time course of smoking withdrawal symptoms. J Abnorm Psychol. 1998 May;107(2):238-51. doi: 10.1037//0021-843x.107.2.238. PMID 9604553
- [Background] Piasecki TM, Niaura R, Shadel WG, Abrams D, Goldstein M, Fiore MC, Baker TB. Smoking withdrawal dynamics in unaided quitters. J Abnorm Psychol. 2000 Feb;109(1):74-86. doi: 10.1037//0021-843x.109.1.74. PMID 10740938
- [Background] Taylor AH, Katomeri M, Ussher M. Acute effects of self-paced walking on urges to smoke during temporary smoking abstinence. Psychopharmacology (Berl). 2005 Aug;181(1):1-7. doi: 10.1007/s00213-005-2216-4. Epub 2005 Oct 15. PMID 15844010
- [Background] Taylor A, Katomeri M. Effects of a brisk walk on blood pressure responses to the Stroop, a speech task and a smoking cue among temporarily abstinent smokers. Psychopharmacology (Berl). 2006 Jan;184(2):247-53. doi: 10.1007/s00213-005-0275-1. Epub 2005 Dec 16. PMID 16362400
- [Background] Taylor AH, Ussher MH, Faulkner G. The acute effects of exercise on cigarette cravings, withdrawal symptoms, affect and smoking behaviour: a systematic review. Addiction. 2007 Apr;102(4):534-43. doi: 10.1111/j.1360-0443.2006.01739.x. PMID 17286639
- [Background] US Department of Health and Human Services: Treating Tobacco Use and Dependence: 2008 Update. A report of the Surgeon General. Public Health Service, Rockville, MD, 2008.
- [Background] Vanderkaay MM, Patterson SM. Nicotine and acute stress: effects of nicotine versus nicotine withdrawal on stress-induced hemoconcentration and cardiovascular reactivity. Biol Psychol. 2006 Feb;71(2):191-201. doi: 10.1016/j.biopsycho.2005.04.006. Epub 2005 Sep 21. PMID 16181727
- [Background] Waters AJ, Shiffman S, Sayette MA, Paty JA, Gwaltney CJ, Balabanis MH. Cue-provoked craving and nicotine replacement therapy in smoking cessation. J Consult Clin Psychol. 2004 Dec;72(6):1136-43. doi: 10.1037/0022-006X.72.6.1136. PMID 15612859
- [Background] Williams MA, Haskell WL, Ades PA, Amsterdam EA, Bittner V, Franklin BA, Gulanick M, Laing ST, Stewart KJ; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Nutrition, Physical Activity, and Metabolism. Resistance exercise in individuals with and without cardiovascular disease: 2007 update: a scientific statement from the American Heart Association Council on Clinical Cardiology and Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2007 Jul 31;116(5):572-84. doi: 10.1161/CIRCULATIONAHA.107.185214. Epub 2007 Jul 16. PMID 17638929
- [Background] Hughes JR. Tobacco withdrawal in self-quitters. J Consult Clin Psychol. 1992 Oct;60(5):689-97. doi: 10.1037//0022-006x.60.5.689. PMID 1401384